CLINICAL TRIAL: NCT02564068
Title: Impact of Oxytocin on Obstructive Sleep Apnea Induced Changes in Sleep
Brief Title: Oxytocin on HR in Sleep Apnea Patient
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Vivek Jain, Principal Investigator, George Washington University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: GWU_IRB_41333
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Results first posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-02

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: All members of the research team except the IP dispensing staff will be blinded for the duration of the research study. Once all the subjects have finished in the research study, and all data is data-locked, the outcomes assessor will then unblind the research data for the statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): These 8 subjects will undergo an "in the sleep-lab" diagnostic polysomnography that would be identical to the one they had for standard of care medical guidelines if they were diagnosed with OSA "in the sleep-lab".
  Interventions: Drug: Oxytocin
- Oxytocin (Experimental): These subjects will undergo another "in the sleep-lab" diagnostic polysomnography that is identical to the one that they had for standard of care to diagnose OSA. Within one hour prior to the research polysomnography the subjects will be given oxytocin (40 IU) intranasally. Outcome measures will be assessed.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — To test that intranasal oxytocin administration blunts the deleterious hypoxia/hypercapnia induced changes in heart rate that occur during nocturnal apnea in patients with OSA, we will examine the changes in heart rate in a group of patients that have recently been diagnosed with OSA. 8 subjects that have recently undergone a standard "in the sleep-lab" diagnostic polysomnography (per standard of care medical guidelines, and not for research purposes) and have been diagnosed with OSA will be recruited into a study to assess the beneficial effects of oxytocin treatment.
  Other Names: Synotocin

SUMMARY:
In human volunteers intranasal administration of oxytocin significantly increases parasympathetic and decreases sympathetic cardiac control. OSA is a very prevalent disease with high cardiovascular risk factors, yet this disease remains very poorly treated. This proposal, based on the current literature and new basic science results detailed above on the role of oxytocin in cardiovascular control, will test if oxytocin administration improves adverse cardiovascular events during the recurrent nocturnal apneas in patients with OSA. This project will lay the groundwork and provide preliminary data to obtain NIH funding to test this important hypotheses more thoroughly and in larger clinical trials.

This study will explore if intranasal oxytocin has any positive cardiovascular benefits in patients with sleep apnea.

DETAILED DESCRIPTION:
Cohort A: 8 Subjects

8 Subjects that have recently undergone either a standard "in the sleep-lab" diagnostic polysomnography or an "at home" PSG test and have been diagnosed with OSA will be recruited into the research study where we will assess the beneficial effects of oxytocin treatment.

These 8 subjects will undergo an "in the sleep-lab" diagnostic polysomnography that would be identical to the one they had for standard of care medical guidelines if they were diagnosed with OSA "in the sleep-lab". This research polysomnography should be performed within 4 weeks of their OSA diagnosis PSG.

These 8 subjects will undergo another "in the sleep-lab" diagnostic polysomnography that is identical to the one that they had for standard of care to diagnose OSA. Within one hour prior to the research polysomnography the subjects will be given oxytocin (40 IU) intranasally. Outcome measures will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Men or women 18 years old or older of any ethnic background
* Subjects that have recently undergone a standard "in the sleep-lab" diagnostic polysonmography (per standard of care medical guidelines), or the "at home" diagnostic test for cohort B, and have been diagnosed with OSA will be recruited into a follow-up study to assess the beneficial effects of oxytocin treatment.

Exclusion Criteria:

* Pregnant or nursing women or women at any child bearing age who are not willing to undergo . methods to prevent pregnancy

  * A female subject of childbearing potential is a nonmenopausal female who has not had a . hysterectomy, bilateral oopherectomy, or medically documented ovarian failure. Menopause . can be assumed to have occurred in a woman when there is either:

    1. Appropriate medical documentation of prior complete bilateral oophorectomy OR
    2. Permanent cessation of previously occurring menses as a result of ovarian failure with . documentation of hormonal deficiency. Ovarian hormonal deficiency is documented by . serum follicle stimulating hormone (FSH) level elevated to within the post-menopausal . . range based on the laboratory reference range where the hormonal assay is performed.
    3. Menopause is defined as occurring 12 months after your last menstrual period and marks the . end of menstrual cycles
* Subjects who are on medications that affect cardiac autonomic function (eg. Beta blockers)
* Smokers
* Subjects who are unable to read or answer questions in the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Jain, MD, Principal Investigator — The George Washington University
Locations (1):
- GW-Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
IPD is not currently planned to be shared with other researchers

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 subjects completed the PSG with intranasal oxytocin administered. There were 8 subjects total.
Groups:
- Oxytocin Only: Subjects will come in for one visit, and will receive only oxytocin
  Oxytocin: To test that intranasal oxytocin administration blunts the deleterious hypoxia/hypercapnia induced changes in heart rate that occur during nocturnal apnea in patients with OSA, we will examine the changes in heart rate in a group of patients that have recently been diagnosed with OSA. Ten subjects that have recently undergone a standard "in the sleep-lab" diagnostic polysomnography (per standard of care medical guidelines, and not for research purposes) and have been diagnosed with OSA will be recruited into a study to assess the beneficial effects of oxytocin treatment.
Period: Overall Study
Arm/Group | Oxytocin Only
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oxytocin
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 43 [36 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8
Body Mass Index (BMI) [Mean (Full Range); unit: (kg)/(m^2)] | 28.3 [23.1 to 39.5]

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Hypopnea Events
Description: Hypopnea events are defined as a reduction in ventilation of 30% that lasted for at least 10 s and resulted in a decrease in arterial saturation of 4% or more. The frequency of hypopnea events is the number of times these events took place during the overnight sleep study.
Time Frame: Duration of single overnight sleep study (variable)
Measure: Mean (Standard Deviation); unit: Incidence of hypopnea events
Arm/Group | Oxytocin
Number analyzed (Participants) | 8
Incidence of hypopnea events | 8.5 (2.0)

2. Primary Outcome: Frequency of Apnea Events
Description: Apnea events are defined as instances of reduction in the peak signal excursion of 90% lasting at least 10 s. Frequency of apnea events is the incidence of these events during a single, over-night sleep study.
Time Frame: Duration of the overnight sleep study (variable)
Measure: Mean (Standard Deviation); unit: Incidence of apnea events
Arm/Group | Oxytocin
Number analyzed (Participants) | 8
Incidence of apnea events | 17.3 (5.7)

ADVERSE EVENTS:
Time Frame: 1 year, 7 months
Arm/Group | Oxytocin Only
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No